CLINICAL TRIAL: NCT05999617
Title: The Effectiveness of Dual Task Exercise Training on Balance, Mobility, Physical Performance and Quality of Life in Children With Cerebral Palsy
Brief Title: Effectiveness of Dual Task Exercise Training in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Fatih Ozden, Assistant Professor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPdualtask
Record Dates: First submitted 2023-08-10; First posted 2023-08-21 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Conventional rehabilitation (stretching, strengthening, balance) plus dual task exercise training (simple math during active stretching, carrying the ball without dropping child while on the balance pad) will be applied 3 days a week for 12 weeks. Interventions will be implemented individually. Patients will be evaluated before and 12 weeks after the interventions.
  Interventions: Other: Rehabilitation
- Control Group (Active Comparator): Conventional rehabilitation program (stretching, strengthening, balance) will be employed.
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — Conventional rehabilitation (stretching, strengthening, balance) and dual task exercise training (simple math during active stretching, carrying the ball without dropping child while on the balance pad) will be applied 3 days a week for 12 weeks. Interventions will be implemented individually. Patients will be evaluated before and 12 weeks after the interventions.

SUMMARY:
Cerebral palsy (CP) is the most common neurological disorder in children and one of the major causes of motor disability. CP causes changes in postural and sensory integration, balance, coordination disorders and muscle weakness due to problems in muscle tone. An effective rehabilitation program is of great importance in solving many problems that can be associated with decreased balance control. Researchers have stated that rehabilitation programs with repetitive special tasks are effective. The aim of the study was to compare the effects of conventional physiotherapy and dual task exercise training in addition to conventional physiotherapy on balance, mobility, physical performance and quality of life in children with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic, monoplegic, unilaterally affected or diplegic children aged 5-12 years with cerebral palsy
* Gross Motor Function Classification (GMFCS) level 1 (walks without restrictions) or 2 (walks with restrictions)
* Understand simple commands
* Signing the consent form

Exclusion Criteria:

* Children and their families who do not want to be involved in the study
* Children with vision and hearing problems
* hildren with secondary orthopedic problems and children with walking aids
* Circumstances that would prevent carrying out assessments and exercise training or communicating

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Pediatric Balance Scale (PBS) | Change from Baseline PBS at 12 weeks
  The scale consists of 14 items measuring parameters such as sitting balance and standing balance. Each item is ranked from 0 to 4. 0 indicates that the instruction cannot be fulfilled, while 4 indicates that it can be fulfilled without any difficulty. The maximum total score is 56.
Timed Up and Go Test (TUG) | Change from Baseline TUG at 12 weeks
  Participants sit in a chair with arms, hips and knees bent approximately 90◦ and feet resting on the floor. Lower limb orthoses are worn if used. Participants are asked to stand up, walk 10 steps, walk around a mark on the floor, walk back to the chair and sit down. The timing of the TUG test starts with the standing movement after the "ready, go" signal and ends when the participants are seated in the chair and the movement is finished.
One Leg Standing Test (OLST) | Change from Baseline OLST at 12 weeks
  Children are tested standing on one leg using their right and left leg respectively. The test is repeated on a hard surface with eyes open and closed. The child is asked to place both hands on the hips and look at a target on the wall at eye level at a distance of 1 meter. The child is asked to stand with one leg while keeping the other leg in a 90 degree flexion position. A stopwatch is used to record the time the child can hold the test position. The examiner ends the test if the child can hold the position for more than 30 seconds and records the elapsed time.
3-Meter Backward Walk Test (3MBWT) | Change from Baseline 3MBWT at 12 weeks
  A distance of 3 m was measured and marked with black tape. Children were asked to follow the black tape with their heels. They were asked to walk backwards quickly with the command 'start'. When the 3 m distance was completed, they were asked to stop. The assessor walked behind the individuals throughout the test.
6 Meter Walk Test (6MWT) | Change from Baseline 6MWT at 12 weeks
  A 6-meter track is determined. Children are asked to walk at a comfortable pace with the command "Start". The stopwatch is stopped by touching the finish line.
The Generic Children's Health-Related Quality of Life Questionnaire (KINDL) | Change from Baseline KINDL at 12 weeks
  The KINDL is a self-report questionnaire available for 3 different age groups: Kiddy-KINDL for children aged 4-7 years, Kid-KINDL for children aged 8-12 years and Kiddo-KINDL for adolescents aged 13-16 years. The total score ranges from 0-100. A higher score represents a better situation.

CONTACTS AND LOCATIONS:
Overall Officials: İsmail Uysal, PhD, Study Director — Muğla Sıtkı Koçman University; Fatih Özden, PhD, Principal Investigator — Muğla Sıtkı Koçman University; İsmet Tümtürk, MSc, Principal Investigator — Süleyman Demirel University; Ahmet İmerci, MD, Principal Investigator — Muğla Sıtkı Koçman University
Locations (1):
- Fethiye Special Son Atilim Special Education and Rehabilitation Center, Muğla, Fethiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No